CLINICAL TRIAL: NCT02216591
Title: Impact of Cognitive Training on Medication Adherence in HIV-infected Individuals
Brief Title: Improving Memory Performance by Applying Cognitive Training
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00053630
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: HIV
Keywords: HIV; Medication Adherence; Working Memory
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Cognitive Training (ACT) (Experimental): The ACT group will complete 12 individual sessions across 6-10 weeks. Sessions will utilize four commercially available memory-training programs from PSSCogRehab 2012, published by Psychological Software Service. The four programs used will be: (1) Sequence recall of digits - auditory (SRD-A), (2) Sequenced Recall Reversed Digits - Auditory (SRRD-A), (3) Sequenced Recall of Words - Visual (SRW-V), and (4) Verbal memory - categorizing (VM-C). In each training session, participants will complete each of the four memory training programs twice.
  Interventions: Device: Active Cognitive Training (ACT)
- Control (CON) (Sham Comparator): The CON group will also complete 12 total sessions across 6-10 weeks. The same four computer programs from PSSCogRehab 2012, published by Psychological Software Service, will be used in the control group sessions. However, the control program will identify the correct responses to participants, such that they do not need to engage their working memory to answer the questions correctly.
  Interventions: Device: Control (CON)

INTERVENTIONS:
Device: Active Cognitive Training (ACT)
  Other Names: PSSCogRehab 2012, published by Psychological Software Service
  Arms: Active Cognitive Training (ACT)
Device: Control (CON)
  Other Names: PSSCogRehab 2012, published by Psychological Software Service
  Arms: Control (CON)

SUMMARY:
The proposed study will test the efficacy of a cognitive training program to improve working memory in a sample of HIV-infected persons. Investigators will assign 40 HIV-infected adults with poor medication adherence to one of two conditions (20/group): the experimental cognitive training intervention or a control training condition. Participants will complete 12 training sessions across 10 weeks and will complete assessments at baseline and post-training. The specific aims are to:

1. Investigate the effects of the cognitive training intervention on working memory and delay discounting in HIV-infected persons.

   Hypothesis 1: Participants assigned to active cognitive training, compared to those in the attention-matched control group, will have greater improvements in working memory and reductions in delay discounting.
2. Characterize adherence to antiretroviral medications in this population and examine medication adherence after cognitive training.

Hypothesis 2: Participants assigned to active cognitive training, compared to those in the attention-matched control group, will have greater improvements in medication adherence.

DETAILED DESCRIPTION:
This study tests the feasibility and preliminary efficacy of a computerized cognitive training program to improve working memory and decrease impulsivity among HIV-infected individuals with poor medication adherence. The specific aims are to: (1) Investigate the effects of the cognitive training intervention on working memory and delay discounting in HIV-infected persons; and (2) Characterize adherence to antiretroviral medications in this population and examine medication adherence after cognitive training.

The research design includes two parts: an eligibility screening and the Cognitive Training study. In Part 1, Eligibility Screening, participants will complete a 2-3 hour battery of standardized measures to assess for study eligibility. Eligible individuals will then be invited to enroll in Part 2, Cognitive Training Study. Part 1 of the study will involved screening approximately 60 participants, with an estimated eligibility rate of 67% for Part 2. In Part 2, participants will be assigned to one of two groups (active cognitive training or control training; 20 participants per group) and will complete 12 training sessions over 10 weeks. Participants assigned to the active cognitive training group will complete computerized modules designed to enhance working memory, while those assigned to the attention-matched control group will complete inactive modules that are not designed to enhance memory. All Part 2 participants will complete assessments at baseline and post-training to evaluate the impact of the training program.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection, diagnosed for > 6 months
* Currently on treatment with antiretroviral medications for > 3 months
* Self-reported medication adherence at less than 90%
* Lives within 15 miles of the research site in stable housing and with no plans to move from the area in the next 3 months

Exclusion Criteria:

* Current substance use disorder
* Any drug use other than alcohol or marijuana in the past year
* Pregnancy
* English non-fluency or illiteracy
* ≤ 8th grade education
* serious neurological disorders, including HIV dementia
* traumatic brain injury
* severe mental illness or acute psychiatric distress
* impaired mental status

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheri L Towe, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Bickel WK, Yi R, Landes RD, Hill PF, Baxter C. Remember the future: working memory training decreases delay discounting among stimulant addicts. Biol Psychiatry. 2011 Feb 1;69(3):260-5. doi: 10.1016/j.biopsych.2010.08.017. Epub 2010 Oct 20. PMID 20965498
- [Background] Lovejoy TI, Suhr JA. The relationship between neuropsychological functioning and HAART adherence in HIV-positive adults: a systematic review. J Behav Med. 2009 Oct;32(5):389-405. doi: 10.1007/s10865-009-9212-9. Epub 2009 Mar 17. PMID 19291386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult persons living with HIV were recruited from the Durham area between January 2015 and May 2016 via flyers and brochures at community-based organizations and infectious diseases clinics.
Pre-assignment Details: Interested persons completed a comprehensive in-person eligibility screen prior to group assignment. 33 participants completed the in-person screen, and 12 were not eligible (5 had no memory impairment, 3 had a current substance use disorder, 2 had a history of brain injury, 1 had severe mental illness, and 1 was not interested).
Groups:
- Active Cognitive Training (ACT): The ACT group will complete 12 individual sessions across 6-10 weeks. Sessions will utilize four commercially available memory-training programs from PSSCogRehab 2012, published by Psychological Software Service. The four programs used will be: (1) Sequence recall of digits - auditory (SRD-A), (2) Sequenced Recall Reversed Digits - Auditory (SRRD-A), (3) Sequenced Recall of Words - Visual (SRW-V), and (4) Verbal memory - categorizing (VM-C). In each training session, participants will complete each of the four memory training programs twice.
  Active Cognitive Training (ACT)
- Control (CON): The CON group will also complete 12 total sessions across 6-10 weeks. The same four computer programs from PSSCogRehab 2012, published by Psychological Software Service, will be used in the control group sessions. However, the control program will identify the correct responses to participants, such that they do not need to engage their working memory to answer the questions correctly.
  Control (CON)
Period: Overall Study
Arm/Group | Active Cognitive Training (ACT) | Control (CON)
Started | 11 | 10
Completed | 11 | 9
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Cognitive Training (ACT) | Control (CON) | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.27 (8.37) | 44.20 (13.01) | 47.90 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Working Memory
Description: Standardized neuropsychological tests of working memory used in this study were the Paced Auditory Serial Addition Task-50 and Neuropsychological Assessment Battery Digits Forward/Digits Backward Test. Using the most up-to-date published normative data, raw test scores were converted to T-scores that corrected for demographic factors such as age and education. T scores can range from 0 to 100, with 50 being average and higher scores indicating better function. The overall working memory score was computed by averaging T-scores of each of the individual tests. To examine intervention effects on working memory outcomes, we conducted a 2 (Arm: ACT vs. CON) × 2 (Time: Baseline vs. Post) mixed-model general linear model analyses. Time was the within-subjects factor defined by baseline versus 10 week follow-up, and study arm was the between-subjects factor. Age and years of education were included as covariates. The means reported here are the mean scores at 10 weeks.
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Error); unit: mean T score on working memory tests
Arm/Group | Active Cognitive Training (ACT) | Control (CON)
Number analyzed (Participants) | 11 | 9
mean T score on working memory tests | 51.33 (2.69) | 43.15 (2.99)
Statistical Analysis 1: Comparison: Active Cognitive Training (ACT) vs Control (CON); Test type: Superiority; p = .013, ANCOVA; Mixed-model general linear model with age and education included as covariates. Time x arm interaction was significant, F(1,16) = 7.76, p = 0.013

2. Secondary Outcome: Change in Delay Discounting
Description: Measured by Monetary-Choice Questionnaire (MCQ), a standardized task that measures delay discounting. Participants are presented with choices between smaller, immediate rewards and larger, delayed rewards (e.g., "Would you prefer $54 today or $80 in 30 days?). Participants' hyperbolic discount parameter (k value) is determined by fitting data to the following discount function equation: Vimmediate = Vdelayed / (1 + kD), in which V is the reward value in dollars and D is delay in days. K-values on this scale can range from 0.00016 to 4.00 and to normalize scores, these values were ranked from 1 to 13 for analyses. A higher rank indicates greater delay discounting.
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: Mean K value rank for MCQ
Arm/Group | Active Cognitive Training (ACT) | Control (CON)
Number analyzed (Participants) | 11 | 9
Mean K value rank for MCQ | 8.62 (1.76) | 8.81 (1.52)
Statistical Analysis 1: Comparison: Active Cognitive Training (ACT) vs Control (CON); Test type: Superiority; p = .274, ANCOVA; Mixed-model general linear model with age and education included as covariates. Time x arm interaction was not significant, F(1,16) = 1.29, p = 0.274

3. Other Pre Specified Outcome: Change in Mean Percent Adherence Across All Antiretroviral Medications
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: Percent of doses
Arm/Group | Active Cognitive Training (ACT) | Control (CON)
Number analyzed (Participants) | 11 | 9
Percent of doses | 94.09 (13.57) | 95.11 (10.20)
Statistical Analysis 1: Comparison: Active Cognitive Training (ACT) vs Control (CON); Test type: Superiority; p = .410, ANCOVA; Mixed-model general linear model with age and education included as covariates. Time x arm interaction was not significant, F(1,16) = .72, p = 0.410

ADVERSE EVENTS:
Time Frame: Approximately 10 weeks (from Baseline to the 10-week assessment)
Arm/Group | Active Cognitive Training (ACT) | Control (CON)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
The overall target sample size of 40 was not reached, and therefore we may have been underpowered to detect differences on secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No